CLINICAL TRIAL: NCT04580069
Title: Effectiveness of Two Rehabilitative Treatments in the Modulation of Inflammation During the Acute Phase in Patients With Knee Prosthesis and Assessment of the Role of the Diet in Determining Post-surgical Inflammation.
Brief Title: Role of Two Rehabilitative Treatments and Diet in the Modulation of Inflammation in Patients With Knee Prosthesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Ospedaliero di Asiago (Other)
Responsible Party: Principal Investigator, Sergio Rigoni, Sergio Rigoni, Presidio Ospedaliero di Asiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POAsiago
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Knee Pain Swelling
Keywords: total Knee Arthroplasty (TKA); C-reactive protein (CRP); erythrosedimentation rate (ESR); Over Knee Oedema (EDO); Under Knee Oedema (EDU); MEDIET Questionnaire
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lymphatic drainage (Experimental): Patients subjected to manual lymphatic drainage
  Interventions: Procedure: Lymphatic drainage
- Connective tissue (Experimental): Patients subjected to connective tissue massage
  Interventions: Procedure: Lymphatic drainage
- control group (Active Comparator): Subjects hat followed standard rehabilitative treatment
  Interventions: Procedure: Lymphatic drainage

INTERVENTIONS:
Procedure: Lymphatic drainage — The interventions follow the validated techniques normally used in international rehabilitation
  Other Names: Connective tissue massage

SUMMARY:
The investigators studied the influence of two aproved rehabilitative treatments, connective tissue techniques and lymphatic drainage, on acute inflammation markers. Furthermore, the role of mediterranean diet on the same values was investigated in the first postoperative period

DETAILED DESCRIPTION:
The main objective of this study is to demonstrate the effectiveness of lymphatic drainage and connective tissue techniques in modulating systemic inflammation. Another objective is to evaluate the existence, at baseline, of a correlation between the inflammation indices and the level of adherence to the Mediterranean diet.

Methods. 34 patients were recruited, and divided into three groups. The control group followed the normal rehabilitation protocol. The other two groups were subjected, in addition to the standard treatment, to manual lymphatic drainage treatment or connective tissue techniques. The outcomes (PCR, ESR, Oedema) were recorded in three stages: upon entering the hospital, 1 week after entry and at follow-up 21 days after surgery.

ELIGIBILITY:
Inclusion criteria

* 50<age<80 years
* Bicompartmental knee arthroplasty
* Weight bearing 7 days after surgery
* Transfusions according to hospital protocol
* Alteration of the indices at T0
* Standard analgesic therapy

Exclusion Criteria:

* Joint replacements from other Units
* Inflammatory arthropathies
* Autoimmune / rheumatic diseases
* Obesity
* Diabetes mellitus
* Infections

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
CRP variation | 21 days
  blood test
ESR variation | 21 days
  blood test
lower limb oedema | 21 days
  leg circumference

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Rigoni, Study Director — Presidio Ospedaliero di Asiago
Locations (2):
- Italy (2):
  - presidio ospedaliero di Asiago, Asiago, Vicenza
  - ULSS 7 Pedemontana, Asiago, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rigoni S, Tagliaro L, Bau D, Scapin M. Effectiveness of two rehabilitation treatments in the modulation of inflammation during the acute phase in patients with knee prostheses and assessment of the role of the diet in determining post-surgical inflammation. J Orthop. 2021 May 15;25:237-243. doi: 10.1016/j.jor.2021.05.016. eCollection 2021 May-Jun. PMID 34099953